CLINICAL TRIAL: NCT06975436
Title: Cobas® BV/CV Test for Use on the Cobas® 5800/6800/8800 Systems: Clinical Performance and Reproducibility
Brief Title: Performance Study of the Cobas® BV/CV Test on Samples From Participants With and Without Symptoms of Bacterial Vaginosis and Candida Vaginitis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Molecular Systems (Unknown)
Responsible Party: Sponsor
Other Study IDs: RD006770
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Bacterial Vaginosis; Candida Vaginitis
MeSH Terms: conditions — Vaginosis, Bacterial; Candidiasis, Vulvovaginal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal swab specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Symptomatic Participants
  Interventions: Diagnostic Test: cobas® BV/CV test; Diagnostic Test: BD Max™ Vaginal Panel; Diagnostic Test: Cepheid Xpert Xpress MVP; Diagnostic Test: Hologic Aptima BV Assay
- Asymptomatic Participants
  Interventions: Diagnostic Test: cobas® BV/CV test

INTERVENTIONS:
Diagnostic Test: cobas® BV/CV test — The cobas® BV/CV test is an automated, qualitative in vitro real-time PCR diagnostic test that detects bacteria and yeast associated with bacterial vaginosis (BV) and candida vaginitis (CV), respectively. The test does not distinguish among the pathogens but can give an overall qualitative result indicating the presence or absence of pathogen(s) associated with BV and/or CV.
Diagnostic Test: BD Max™ Vaginal Panel — This is an FDA-cleared diagnostic test that will be used as labelled. It will serve as one of three comparators in this study for determining BV patient infection status.
  Groups: Symptomatic Participants
Diagnostic Test: Cepheid Xpert Xpress MVP — This is an FDA-cleared diagnostic test that will be used as labelled. It will serve as one of three comparators in this study for determining BV patient infection status.
  Groups: Symptomatic Participants
Diagnostic Test: Hologic Aptima BV Assay — This is an FDA-cleared diagnostic test that will be used as labelled. It will serve as one of three comparators in this study for determining BV patient infection status.
  Groups: Symptomatic Participants

SUMMARY:
In the clinical performance part of this study, prospectively acquired clinician-collected and clinician-instructed, self-collected vaginal swab specimens collected in cobas® PCR Media will be taken from a minimum of 500 symptomatic individuals with a clinical presentation consistent with vaginitis, vaginosis, or both. Additionally, a minimum of 100 asymptomatic individuals will also be enrolled in the study. The cobas® BV/CV assay amplifies and detects the deoxyribonucleic acid (DNA) of pathogens associated with bacterial vaginosis (BV) and candida vaginitis (CV). The BV results will be compared with the patient infection status (PIS) established by using 3 Food and Drug Administration (FDA)-cleared commercial assays, and the CV results will be compared with the PIS established with the use of culture plus MALDI-TOF (matrix-assisted laser desorption/ionization time-of-flight).

The primary objective of the clinical performance study is to evaluate the performance (sensitivity and specificity) of cobas® BV/CV to determine the presence of BV and/or CV in the intended use patient population when being tested on cobas® 6800/8800 systems. The secondary objective is to evaluate the equivalency of cobas® BV/CV between the cobas® 5800 system and cobas® 6800/8800 systems.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Symptomatic Participants:

* Symptomatic participants with a clinical presentation consistent with vaginitis, vaginosis, or both; symptoms may include abnormal vaginal discharge, painful or frequent urination, vaginal itching or burning or irritation, painful or uncomfortable intercourse, and/or abnormal vaginal odor.
* Participants aged 14 years or older who are willing and able to provide written, informed consent; for pediatric participants, written assent and parent/legal guardian consent, as applicable by the institutional review board/ethics committee (IRB/EC).

Inclusion Criteria for Asymptomatic Participants:

* Apparently healthy participants aged 14 years or older who are willing and able to provide written, informed consent; for pediatric participants, written assent and parent/legal guardian consent, as applicable by the IRB/EC.

Exclusion Criteria:

Exclusion Criteria for Symptomatic Participants:

* Participants not meeting the above described inclusion criteria will be excluded from the study.
* Use of any azole-containing antimicrobial (oral or vaginal) within the 7 days prior to study enrollment.
* Prior enrollment in this study.
* Use of any lubricants (eg, Replens, RepHresh) within 3 days prior to sample collection
* Use of douches, vaginal deodorizers, or other intravaginal products within 3 days prior to sample collection. The use of tampons or pads during menses should not be considered exclusionary criteria.
* Contraindication to vaginal swab sampling.
* Asymptomatic participants who do not have any signs or symptoms consistent with vaginitis, vaginosis, or both, as described above.

Exclusion Criteria for Asymptomatic Participants:

* Prior enrollment in this study.
* Participants with a clinical presentation consistent with vaginitis, vaginosis, or both; symptoms may include abnormal vaginal discharge, painful or frequent urination, vaginal itching or burning or irritation, painful or uncomfortable intercourse, and/or abnormal vaginal odor.

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The intended use population will be a minimum of 500 symptomatic participants with a clinical presentation consistent with vaginitis, vaginosis, or both. A population of a minimum of 100 asymptomatic participants will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 738 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Clinical Sensitivity of the cobas® BV/CV Test on the cobas® 6800/8800 Systems for Detecting the Presence of BV and/or CV Compared with the Patient Infection Status | Day 1
  The sensitivity of a diagnostic test is the percentage of true positive (TP) tests out of all patients with a condition. It is calculated as follows: 100% x (TP)/(TP + false negatives (FN)). The BV test results will be compared with the patient infection status (PIS) established by using 3 Food and Drug Administration (FDA)-cleared commercial assays. The CV test results will be compared with the PIS established by using selective culture and MALDI-TOF.
Clinical Specificity of the cobas® BV/CV Test on the cobas® 6800/8800 Systems for Detecting the Presence of BV and/or CV Compared with the Patient Infection Status | Day 1
  The specificity of a diagnostic test is the percentage of true negative (TN) tests out of all patients who do not have a condition. It is calculated as follows: 100% x (TN)/(TN + false positives (FP)). The BV test results will be compared with the patient infection status (PIS) established by using 3 FDA-cleared commercial assays. The CV test results will be compared with the PIS established by using selective culture and MALDI-TOF.
Positive Predictive Value of the cobas® BV/CV Test on the cobas® 6800/8800 Systems for Detecting the Presence of BV and/or CV Compared with the Patient Infection Status | Day 1
  The positive predictive value of a diagnostic test is the percentage of true positive (TP) tests out of all of the positive findings. It is calculated as follows: 100% x (TP)/(TP + FP). The BV test results will be compared with the patient infection status (PIS) established by using 3 FDA-cleared commercial assays. The CV test results will be compared with the PIS established by using selective culture and MALDI-TOF.
Negative Predictive Value of the cobas® BV/CV Test on the cobas® 6800/8800 Systems for Detecting the Presence of BV and/or CV Compared with the Patient Infection Status | Day 1
  The negative predictive value of a diagnostic test is the percentage of true negative (TN) tests out of all of the negative findings. It is calculated as follows: 100% x (TN)/(TN + FN). The BV test results will be compared with the patient infection status (PIS) established by using 3 FDA-cleared commercial assays. The CV test results will be compared with the PIS established by using selective culture and MALDI-TOF.

SECONDARY OUTCOMES:
Equivalency of the cobas® 5800 System and the cobas® 6800/8800 Systems: Clinical Sensitivity of the cobas® BV/CV Test for Detecting the Presence of BV and/or CV | Day 1
  The sensitivity of a diagnostic test is the percentage of true positive (TP) tests out of all patients with a condition. It is calculated as follows: 100% x (TP)/(TP + false negatives (FN)). The BV test results obtained with each cobas® system will be compared with the patient infection status (PIS) established by using 3 FDA-cleared commercial assays. The CV test results obtained with each cobas® system will be compared with the PIS established by using selective culture and MALDI-TOF.
Equivalency Between the cobas® 5800 System and the cobas® 6800/8800 Systems: Clinical Specificity of the cobas® BV/CV Test for Detecting the Presence of BV and/or CV | Day 1
  The specificity of a diagnostic test is the percentage of true negative (TN) tests out of all patients who do not have a condition. It is calculated as follows: 100% x (TN)/(TN + false positives (FP)). The BV test results obtained with each cobas® system will be compared with the patient infection status (PIS) established by using 3 FDA-cleared commercial assays. The CV test results obtained with each cobas® system will be compared with the PIS established by using selective culture and MALDI-TOF.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (8):
  - Matrix Clinical Research, Los Angeles, California
  - M3 Wake Research - San Diego at Convoy, San Diego, California
  - Red Rocks OBGYN, Lakewood, Colorado
  - Altus Research, Lake Worth, Florida
  - Washington University, St Louis, Missouri
  - Eastern Carolina Women's Center, New Bern, North Carolina
  - Unified Women's Clinical Research/Lyndhurst, Winston-Salem, North Carolina
  - Planned Parenthood Gulf Coast, Houston, Texas
- Diagnostic Consultative Center "Ascendent" Ltd., Sofia, Bulgaria
- Centre Hospitalier Universitaire Vaudois (Chuv), Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No